CLINICAL TRIAL: NCT05357573
Title: An Open-Label, Multi Center, Single-Cohort, Post-Marketing Phase 4 Study to Evaluate the Efficacy, Pharmacodynamics, and Safety of the Anti-FGF23 Antibody, KRN23, in Adult Chinese Patients With Tumor-Induced Osteomalacia (TIO)
Brief Title: Study to Assess the Safety, Pharmacokinetics and Efficacy of KRN23 in Adult Chinese Patients With TIO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN23-CN007
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Tumor-Induced Osteomalacia (TIO)
MeSH Terms: conditions — Oncogenic osteomalacia | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KRN23 (Experimental): KRN23 administered subcutaneously (SC) every 4 weeks for 48 weeks. The dose varies according to serum phosphorus level which include 0.3,0.6,1.0,1.4 and 2.0 mg/kg.
  Interventions: Drug: KRN23

INTERVENTIONS:
Drug: KRN23 — KRN23 is a sterile clear colourless and preservative free solution supplied in single use 5 mL vials containing 1 mL of KRN23 at a concentration of 30mg/mL
  Other Names: Burosumab; Crysvita

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics and efficacy of KRN23 in adult Chinese patients with TIO

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of TIO based on evidence of excessive FGF23 that is not amenable to cure by surgical excision of the offending tumor (documented by Investigator)
2. Male or female Chinese patients aged ≥18 years at the time of signing the informed consent form
3. Have a fasting serum phosphorus level < 2.5 mg/dL (0.81 mmol/L) at Screening
4. Have a serum iFGF23 level ≥ 100 pg/mL by Kainos assay at Screening
5. Have a TmP/GFR < 2.5 mg/dL at Screening
6. Have an estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73m2(using CKD-EPI formula) at Screening. Subjects with an eGFR ≥ 30 but < 60 mL/min at screening will be considered eligible so long as in the opinion of the Investigator the decline in renal function is not related to nephrocalcinosis
7. Have a corrected serum calcium level < 10.8 mg/dL (2.69 mmol/L) at Screening (Corrected serum calcium = serum calcium in mg/dL + 0.8 × [4 - serum albumin in g/dL])
8. Have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study (female patients of child-bearing potential only)
9. Be willing to use an effective method of contraception while participating in the study (sexually active patients of child bearing potential) and for 12 weeks after last dose of study drug. Women of non child bearing potential are defined as permanently sterile (i.e. due to hysterectomy or bilateral oophorectomy) or postmenopausal (defined as at least 12 months postcessation of menses without an alternative medical cause). Postmenopausal status of female patients will be confirmed with a Screening serum follicle stimulating hormone (FSH) level >40 mIU/mL
10. Be willing to provide access to prior medical records to determine eligibility including imaging, biochemical, and diagnostic, medical, and surgical history data
11. Provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures
12. Be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments (in the opinion of the Investigator)

Exclusion Criteria:

1. Use of the following drugs within 14 days prior to screening: pharmacologic vitamin D metabolites or analogs, or drugs for treating TIO including oral phosphate, aluminum hydroxide antacids, acetazolamide, or thiazide diuretics
2. Medication to suppress parathyroid hormone (PTH) (e.g., cinacalcet hydrochloride) within 60 days prior to screening
3. Blood or blood product transfusion within 60 days prior to screening
4. History of malignancy within 5 years of study entry with the exception of PMT-MCT (phosphaturic mesenchymal tumors of the mixed connective tissue type)
5. Positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibody at Screening, or prior history of positive test
6. Predisposition to infection, or history of recurrent infection or known immunodeficiency
7. Pregnant or breastfeeding at screening or intention to become pregnant during the study; for male subjects, the partner's intention to become pregnant during the study
8. Use of an investigational product (IP) or device within 4 months prior to screening, or planning to receive other IP before completing all assessments in this study.
9. Use of KRN23, or any other therapeutic mAb within 90 days before signing the informed consent form.
10. History of allergic or anaphylactic reactions to KRN23, any of the KRN23 ingredients, or any other monoclonal antibodies
11. Anyone otherwise considered unsuitable participation in the study by the investigator or subinvestigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in mean serum phosphorus level at the end of the dosing cycle. | Week 20, 24, 28, 32, 36, 40, 44 and 48

SECONDARY OUTCOMES:
Change from Baseline in mean serum phosphorus level. | Week 22
Proportion of patients achieving serum phosphorus level above the lower limit of normal (LLN; 2.5 mg/dL [0.81 mmol/L]) | Week 22
Proportion of patients achieving mean serum phosphorus level above the LLN (2.5 mg/dL [0.81 mmol/L]) at the end of the dose cycle as averaged across dose period | Weeks 20, 24, 28, 32, 36, 40, 44 and 48
Change from Baseline in mean level of serum 1,25(OH)2D over time | Week 0, 1, 2, 12, 16, 24, 36 and 48
Change from Baseline in mean level of serum creatinine over time | Week 0, 4, 8, 12, 16, 24, 36 and 48
Change from Baseline in mean level of urinary phosphorus over time | Week 0, 4, 8, 12, 16, 24, 36 and 48
Change from Baseline in level of tubular reabsorption of phosphate(TRP) over time | Week 0, 4, 8, 12, 16, 24, 36 and 48
Change from Baseline in ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR) over time | Week 0, 4, 8, 12, 16, 24, 36 and 48
Change in concentration of alkaline phosphatase (ALP) over time | Week 0, 8, 16, 24 and 48
Change in concentration of bone-specific alkaline phosphatase (BALP) over time | Week 0, 8, 16, 24 and 48
Change in concentration of carboxy-terminal cross-linked telopeptide of type 1 collagen (CTx) over time | Week 0, 8, 16, 24 and 48
Change in concentration of procollagen type 1 N propeptide(P1NP) over time | Week 0, 8, 16, 24 and 48
Change in concentration of osteocalcin (OC) over time | Week 0, 8, 16, 24 and 48
Change from Baseline in six-minute walking test (6MWT) over time | Week 0, 12, 24 and 48
  This test will measure the distance that the subject can walk a previously measured course in a period of 6 minutes.
Change from Baseline in Brief Pain Inventory (BPI) score over time | Week 0, 12, 24 and 48
  Evaluate the degree of pain and its impact on daily functioning over previous 24 hours, the subject will fill out a 15-item self-administered questionnaire. The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). The severity of pain in the last 24 hours is rated on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
Change from Baseline in Brief Fatigue Inventory (BFI) score over time | Week 0, 12, 24 and 48
  Evaluate the degree of fatigue and its impact on daily functioning over previous 24 hours, the subject will fill out a 9-item self-administered questionnaire.
  Two dimensions are measured: fatigue severity (now, usual and worst) and the impact of fatigue on functioning (fatigue interference with general activity, mood, walking ability, normal work, relations with other people, enjoyment of life). The severity of fatigue in the last 24 hours is rated on a scale of 0 (no fatigue or does not interfere) to 10 (fatigue as bad as you can imagine or completely interferes). Scores are normalized to a 0-10 metric where 0 was the best health state and 90 was the worst.
36-item short-form health survey (SF-36) scores to examine health-related Quality of Life | Week 0, 12, 24 and 48
  Evaluate physical and mental health status, the subject will fill out a 36-item self-administered questionnaire.
  The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). The score will be calculated based on scoring system, and the Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.

OTHER OUTCOMES:
Change from Baseline in bone mineral density over time | Week 0, 24 and 48
Radiologic healing or resolution of pre-existing fractures and/or pseudofractures, as defined by skeletal survey at Baseline and subsequent targeted radiography. | Week 0, 12, 24, 36 and 48
Radiologic healing or resolution of pre-existing fractures and/or pseudofractures, as defined by skeletal survey at Baseline and 99mTc-labelled bone scan | Week 0, 24 and 48
Safety of KRN23 by studying the number of Adverse Events (including laboratory and imaging assessments) | Week 0 to Week 48
  Incidence and frequency of AEs and SAEs, including clinically significant changes in laboratory assessments as well as ECHO, ECG, ultrasound, vital sign, tumor images and Anti-KRN23 antibody.
Safety of KRN23 by studying the severity of Adverse Events (including laboratory and imaging assessments) | Week 0 to Week 48
  Severity of AEs and SAEs, including clinically significant changes in laboratory assessments as well as ECHO, ECG, ultrasound, vital sign, tumor images and Anti-KRN23 antibody.
Safety of KRN23 by studying the relatedness of Adverse Events (including laboratory and imaging assessments) | Week 0 to Week 48
  Relatedness between KRN23 and AEs/SAEs, including clinically significant changes in laboratory assessments as well as ECHO, ECG, ultrasound, vital sign, tumor images and Anti-KRN23 antibody.
Pharmacokinetics: KRN23 concentrations | Week 0, 1, 2, 4, 16, 20, 22, 24 and 48
  KRN23 concentration in the Mid and end of dose cycles.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Shanghai Jiaotong University Affiliated Sixth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No